CLINICAL TRIAL: NCT00708734
Title: Exercise Intervention to Reduce Postural Instability in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F5070-R
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis
Keywords: exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): functional exercise training
  Interventions: Behavioral: functional exercise training

INTERVENTIONS:
Behavioral: functional exercise training — twice weekly group sessions for 5 weeks

SUMMARY:
This is a one year pilot study evaluating the feasibility of a 10 week, twice weekly, group functional exercise sessions in individuals with knee osteoarthritis and its effect on gait and balance measures.

DETAILED DESCRIPTION:
Impaired gait and balance (referred to as impaired postural stability) is one of the most significant causes and consequences of falls. Persons with osteoarthritis (OA) of the knee represent one of the largest patient populations with impaired postural stability. Specifically, knee OA has been shown to reduce walking speed, shorten stride length and prolong the stance phase of the gait cycle. Patients with knee OA also have less range of motion of the hip, knee and ankle joints. Functional Exercise Training (FET) has been shown to improve gait and balance, and decrease falls and associated fall-related injuries in the general elderly populations. While traditional exercise programs have not been well-tolerated in persons with knee OA (due to pain), we are interested in whether a tailored FET intervention would be effective in this patient population. Immediate Objectives: O1: Characterize the etiology and mechanisms of postural instability in persons with knee OA; O2: Refine the clinical protocol for FET in veterans with knee OA; O3: Refine the sampling plan; O4: Refine the data collection protocol. This 1-year feasibility study uses a prospective cohort design, including data collection at baseline and three points post intervention (10 weeks {end of intervention}, 15 weeks, and 20 weeks). Subjects with knee osteoarthritis are enrolled. Inclusion Criteria: Age 60 and older; Corrected vision not worse than 20/50; Ability to ambulate household distances without an assistive device - minimum functional status for ambulation as primary mode of mobility; presence of knee OA based on clinical and radiological criteria. Sample size: 36 subjects. Intervention: Participants attend FET class twice weekly for 10 weeks. Our primary outcome is a composite measures of postural stability (gait and balance) and OA symptoms/physical disability. Secondary outcome measures include fall self-efficacy and quality of life. We also collect case histories on postural instability and falls as well as data on key mediating variables, including level of participation (dose of intervention), body mass index (BMI), analgesic use, tolerance of intervention, and number of joints affected by OA. Measurement tools: Balance is measured with Sensory Organization Test and Limits of Stability test using Neurocom Smart Balance Master and Berg Balance Test; Gait is measured with multiple kinetic and kinematic variables using VICON 3-D Motion Analysis System; OA symptoms/physical disability are measured using Western Ontario and McMaster University Arthritis Index (WOMAC) Osteoarthritis Index; Fall self-efficacy by Modified Fall Self Efficacy Scale; and Quality of life by Short Form 36v (SF-36v).

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older.
* Corrected vision not worse than 20/50.
* Ability to ambulate household distances without an assistive device - minimum functional status for ambulation as primary mode of mobility.
* Presence of knee OA based on clinical and radiological criteria.

Exclusion Criteria:

* Cognitive impairment with Mini Mental State Exam (MMSE) score <24; Scores at or below 24 indicate cognitive impairments, limiting ability to participate in the group and/or remember instructions.
* Metastatic cancer, since this limits ability to fully participate in the group and/or complete the intervention due to limited life expectancy and changing functional status.
* Central or peripheral neurological dysfunction e.g. diagnosis of hemiparesis, cerebellar dysfunction, Parkinson's disease , peripheral neuropathy with or without foot drop, as determined by medical record review and physical exam; Severe Peripheral Vascular Disease with claudication or Spinal Stenosis with pseudoclaudication/chronic low back pain; These impairments would further impair gait and balance, and would jeopardize safety during the intervention and/or confound the effect of the intervention.
* Lower extremity amputations, or foot deformities; Mobility limitations due to altered lower extremity skin integrity/ulcer, where weight-bearing would be contraindicated (foot ulcers), since this would affect gait and balance measures.
* Use of medications known to impair balance, e.g. antipsychotics, benzodiazepines, anti-epileptics, etc. which would affect gait and balance measures.
* Severe arthritis limiting basic activities of daily living (ADL) and were offered or are pending joint replacement, since it is unlikely that any non-pharmacological intervention would be effective.
* Total knee replacement on one or both sides, since gait and balance changes due to total knee replacement would confound the effect of interventions.
* Current involvement in physical therapy, since it would confound results.
* Medically unstable upon exam, i.e. poorly controlled blood pressure or blood sugar, unstable coronary artery disease, since group participation may compromise medical status.
* Morbid obesity (BMI>40) due to potential changes in gait variables (speed, cadence, stride length).
* Weight over 300 pounds (due to limitations of Neurocom force plate).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Bulat, MD, Principal Investigator — James A. Haley Veterans' Hospital
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: functional exercise training
  functional exercise training: twice weekly group sessions for 10 weeks This one year feasibility study had a planned sample of 35 subjects. Of the 94 subjects that were screened, 45 did not meet criteria, and 39 declined participation after screening. Of the ten subjects enrolled, three completed the intervention and follow up sessions. The remaining seven were unable to continue participation after enrollment due to a number or reasons including vertigo, moving out of state, total knee replacement after baseline, unable to contact, scheduling conflicts, and a fall with fracture, precluding weight-bearing exercise.
Period: Overall Study
Arm/Group | Arm 1
Started | 10 (94 subjects were screened, 45 did not meet criteria, and 39 declined participation after screening.)
Completed | 3 (Ten subjects enrolled, three completed the intervention and all follow up sessions.)
Not Completed | 7
Not completed — scheduling conflict | 2
Not completed — moved | 1
Not completed — leg injury | 1
Not completed — knee replacement | 1
Not completed — vertigo | 1
Not completed — leg fracture | 1

BASELINE CHARACTERISTICS:
Population: age over 50 and gender
Groups:
- Functional Exercise Training: functional exercise training
  functional exercise training: twice weekly group sessions for 5 weeks
Arm/Group | Functional Exercise Training
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] — Age criteria for participants in the study was age 50 and older.
  years | 66.5 [50 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participants in the study
  Participants
    Female | 1
    Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Gait and Balance Measures
Description: Assessment of balance using the (sensory organization test, limits of stability, berg balance) and gait using 3D motion capture.
Time Frame: 5 months
Population: The purpose of this pilot study was to evaluate the feasibilty of a structured, group exercise program in this population. Only 3 of 10 participants completed the study, due to high attrition, the project was considered unfeasible and data was not analysis.
Groups:
- Composite Measures of Gait and Balance: Measurement of gait and balance using standardized tools
Arm/Group | Composite Measures of Gait and Balance
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date was collected from date of participant enrollment through the close of the study
Groups:
- Functional Exercise Training: functional exercise training
  functional exercise training: twice weekly group sessions for 10 weeks This one year feasibility study had a planned sample of 35 subjects. Of the 94 subjects that were screened, 45 did not meet criteria, and 39 declined participation after screening. Of the ten subjects enrolled, three completed the intervention and follow up sessions. The remaining seven were unable to continue participation after enrollment due to a number or reasons including vertigo, moving out of state, total knee replacement after baseline, unable to contact, scheduling conflicts, and a fall with fracture, precluding weight-bearing exercise.
Arm/Group | Functional Exercise Training
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No